CLINICAL TRIAL: NCT06218667
Title: CHARIOT: a Phase 1b/2 Study of Androgen Deprivation Therapy and Copanlisib in High-Risk Localized Prostate Cancer Patients Prior to Radical Prostatectomy
Brief Title: A Study of Copanlisib in Combination with Degarelix in People with Prostate Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study drug not available per sponsor
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-331
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: Androgen Deprivation Therapy; Copanlisib; Radical Prostatectomy; Degarelix
MeSH Terms: conditions — Prostatic Neoplasms | interventions — copanlisib; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Copanlisib in Combination With Degarelix (Experimental): Phase 1b: The starting Dose level 1 will be 45 mg with the intent of dose escalating to the standard dose of 60 mg approved for heme malignancy. In the event of > =2 DLT at Dose level 1 (45 mg) the study will be terminated. If >= 2 DLT in patients at Dose level 2 (60 mg), Dose level 1 (45 mg) will be the RP2D if <= 1 DLT out of 6 patients at this dose.
  Phase 2: Patients may dose reduce at the discretion of the investigator to the lowest dose of 45 mg. Participants who do not tolerate the copanlisib dose of 45 mg must discontinue study treatment permanently.
  Interventions: Drug: Copanlisib; Drug: Degarelix; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Copanlisib — Dose level 1 (starting dose): 45 mg of copanlisib IV weekly x 3 weeks on/1 week off Dose level 2 (standard dose): 60 mg of copanlisib IV weekly x 3 weeks on/1 week off
Drug: Degarelix — Degarelix (GnRH antagonist): 240 mg loading dose sub-cutaneous once on C1D1; 80 mg maintenance dose on C2D1 and C3D1.
Procedure: Radical Prostatectomy — Standard treatment

SUMMARY:
The researchers are doing this study to find out whether copanlisib in combination with degarelix, given before standard surgical treatment (radical prostatectomy), is a safe and effective treatment that causes few or mild side effects for people who have localized high-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and privacy authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.
* Individuals with prostate cancer 18 years of age and above
* Histological or cytological evidence of prostate cancer
* Documented high-risk localized prostate cancer based on one or more of the following NCCN criteria:

  1. PSA >20ng/ml or
  2. Gleason ≥8 or
  3. Clinical stage ≥cT3a
* Known PTEN status:

  1. PTEN loss by IHC for participants in the PTEN loss cohort
  2. PTEN intact by IHC for participants in the exploratory PTEN intact cohort (only available if PTEN intact cohort is opened)
* Candidate for RP as determined by treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Appendix A: Performance Status Criteria)
* Normal organ function with acceptable initial laboratory values within 28 days of registration:

  * ANC ≥ 1.5 K/mcL
  * Hemoglobin ≥ 9g/dL
  * Platelet count ≤100 K/mcL
  * Creatinine ≤ 1.5 x the institutional upper limit of normal (ULN)
  * Potassium within institutional normal range
  * Total Bilirubin ≤ 1.5 x ULN (Note: In participants with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, participant may be eligible)
  * SGOT (AST) ≤ 2.5 x ULN
  * SGPT (ALT) ≤ 2.5 x ULN
  * GFR (MDRD) ≥ 30 mL/min/1.73 m^2
* Participants must agree to use a medically acceptable method of birth control (i.e., spermicide in conjunction with a barrier such as a condom) or sexual abstinence prior to registration, for the duration of study participation and for at least 5 months after the last treatment with copanlisib.

Exclusion Criteria:

* Radiographic evidence of distant (extra-pelvic) metastatic prostate cancer on CT and/or MRI, bone scan or PET scan
* On ADT (GnRH agonists or antagonists) for > 4 weeks at time of consent
* Prior radiation to prostate
* Medical conditions such as uncontrolled hypertension or cardiac disease that would, in the opinion of the investigator preclude participation in this protocol
* A diagnosis of diabetes (type 1 or 2) on medications for the purpose of treating hyperglycemia or HgbA1C > 7 will be excluded from study
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for basal or squamous cell skin cancer or superficial bladder cancer that has previously been treated.
* Use of any prohibited concomitant medications including herbal supplements Medications With the Potential for Drug-Drug Interactions) within 2 weeks prior to treatment start
* Receiving any other investigational agents within 4 weeks or 5x the half-life of investigational agent (whichever is longer) from this study's treatment start
* Known allergy to any of the compounds under investigation
* Any other condition which, in the opinion of the Investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 0 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
phase Ib determine the recommended phase 2 dose (RP2D) of copanlisib in combination with degarelix | 1 year
  DLTs are any of the following events not clearly due to the underlying disease or extraneous causes. Toxicities will be evaluated using CTCAE version 5.0 (CTCAE v5.0). Only toxicities that meet DLT definitions within the DLT assessment window (one 28-day cycle) and are attributed to degarelix, copanlisib or copanlisib plus degarelix will be counted as DLTs.
Phase 2 determine the rate of pCR or MRD at Radical Prostatectomy | 2 years
  pCR will be defined as the absence of morphologically identifiable carcinoma in the RP specimen. MRD will be defined as ≤ 5mm of residual tumor in the RP specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm